CLINICAL TRIAL: NCT03254472
Title: Defining Use and Misuse of BIoMarkers Dosage and Trends in Observed Concentration Over Time: a BIg Data Analysis
Brief Title: Big Data Analysis of the Use of bIomarkers Concentration
Acronym: rUBIDIuM
Status: Completed | Type: Observational
Sponsor: Hospital Avicenne (Other)
Collaborators: Roche Diagnostics GmbH (Industry); ProBayes (Unknown); Biorance Laboratoires Réunis (Unknown)
Responsible Party: Principal Investigator, Christophe Meune, MD-PhD, Professor, Hospital Avicenne
Other Study IDs: 2017-003438-10
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Biological Markers; Inappropriate Prescribing
Keywords: Biological markers; Professional practice; Big data analysis; Measured concentrations; Cardiac markers; Troponin; NTproBNP; Creatinin; INR; Hemogram; Lipid profile

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measured concentrations of biomarkers

SUMMARY:
The investigators conducted a retrospective analysis of all measured concentrations performed in a large subset of laboratories located in the French Brittany from February 2010 the 17th to August 2015 the 30th, in adults over 20 years old.

The investigators are aimed at studying physicians' use and eventually misuse of biomarkers dosage and the characteristics of a broad population based on some biomarkers concentrations.

DETAILED DESCRIPTION:
The rUBIDIuM study is a retrospective analysis that included all tests (but not including DNA analysis or HIV tests) performed in a large subset of laboratories located in the French Brittany from February 2010 the 17th to August 2015 the 30th. The area of study covers most of the Ille-et-Vilaine and a part of the Côtes d'Armor department in Brittany. The respective surface of these departments is 6775 and 6878 km2. All labs belong to the Biorance Laboratory group (consortium of 33 labs, Biorance Laboratoires Réunis) and are equipped with Roche Diagnostics instruments (Elecsys2010® analyzer, Roche diagnostics, Meylan, France).

The main objectives are to study physicians' use and eventually misuse of biomarkers dosage and the characteristics of this broad population based on some biomarkers concentrations.

For all adult patients >20y that came to a participating lab during the study period, the investigators collected the following information: demographics data, data about the prescription (date of order, list of analysis recommended, the date of blood collection and analysis), about the prescribers and the results of the analyses. After a de-identifying process, data were aggregated.

the initial analyses will 1) examine the biological tests (number, types…) ordered in a large cohort of patients, in the total population and the subgroups based on gender, age, time period, kind of lab and physicians' specialty, 2) examine the results/concentration of the analyses: blood chemistry, creatinin concentration, cardiac enzymes, natriuretic peptides, INR, lipid profile, hemogram…

ELIGIBILITY:
Inclusion Criteria:

* All adult patients >20 that came to a participating lab (Biorance Laboratoires Réunis) during the study period for biological measurement

Exclusion Criteria:

* DNA analysis, HIV test

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort that included all analyses performed in a large subset of laboratories located in the French Brittany from February 2010 the 17th to August 2015 the 30th.
  The extract data corresponded to 74,502,510 analyses performed in 585,745 distinct adult patients >20y
Sampling Method: Non-Probability Sample
Enrollment: 585745 (Actual)
Dates: Start 2010-02-17 (Actual); Primary Completion 2015-08-30 (Actual); Study Completion 2015-09-10 (Actual)

PRIMARY OUTCOMES:
biomarker dosage prescription | August 2017
  physicians' use and eventually misuse of biomarkers dosage

SECONDARY OUTCOMES:
Biomarkers dosage numbers | August 2017
  Biomarkers dosage numbers before and after new treatments, released of guidelines, new tests...
Biomarkers in geriatric patients | August 2017
  biomarkers dosages and concentration in elderly/very elderly patients
Population's characteristics | August 2017
  physicians' use and eventually misuse of biomarkers dosage

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Meune, MD PhD, Principal Investigator — Avicenne Hospital
Locations (1):
- Avicenne Hospital, Bobigny, France

IPD SHARING:
Plan to Share IPD: No
Only aggregated data are available